CLINICAL TRIAL: NCT03289403
Title: The Role of Immunomodulatory Treatment in Success of ICSI in Patients Who Have Infertility With Autoimmune Thyroiditis
Brief Title: The Role of Immunomodulatory Treatment in Success of ICSI in Patients With Autoimmune Thyroiditis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICSI/ Autoimmune thyroiditis
Record Dates: First submitted 2017-09-17; First posted 2017-09-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Infertility; Autoimmune Thyroiditis
MeSH Terms: conditions — Infertility; Thyroiditis, Autoimmune | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Patients will receive thyroxine , low dose aspirin , low dose selenium, Calcium and vitamin D and immunomodulatory drugs(prednisolone, hydroxychloroquine, azathioprin, IV immunoglobulins)
  Interventions: Drug: Immunomodulatory
- Control group (Active Comparator): Patients will receive thyroxine , low dose aspirin , low dose selenium, Calcium and vitamin D.
  Interventions: Drug: Thyroxine

INTERVENTIONS:
Drug: Immunomodulatory — Patients will receive thyroxine , low dose aspirin , low dose selenium, Calcium and vitamin D before ICSI cycle.
  Moreover, patients will receive a treatment course of immunomodulatory drugs for 3 -6 months before ICSI cycle:
  1. Prednisnlone 40mg for 2 weeks to be lowered gradually till become 5mg after 6 weeks and to be continued
  2. Hydroxychloroquine according to body weight, patients who develop hypersensitivity will be shifted to Azathioprin.
  3. Immunoglobulins will be used in cases not responding to treatment.
  Arms: Study group
Drug: Thyroxine — Patients will receive thyroxine , low dose aspirin , low dose selenium, Calcium and vitamin D before ICSI cycle.
  Patients will not receive immunomodulatory drugs
  Arms: Control group

SUMMARY:
The aim of the work is to determine whether the use of immunomodulatory drugs could improve the reproductive of outcome of infertile patients who have autoimmune thyroiditis with positive autoimmune antibodies undergoing IVF-ET.

ELIGIBILITY:
Inclusion Criteria:

* Infertility patients who have autoimmune thyroiditis With positive autoimmune thyroiditis and TSH level above 2 IU.

Exclusion Criteria:

* All patients who have other autoimmune diseases especially antiphospholipid syndrome, hepatitis c viral disease.

Patients who have any medical disorders ( eg. D.M. HTN .Epilepsy ….)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 194 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
The Number of Participants Who Achieved clinical Pregnancy | 6 weeks after embryo transfer

SECONDARY OUTCOMES:
The Number of Participants Who Achieved Ongoing Pregnancy | 18 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Sayed, Prof., Study Chair — Aljazeera (Al Gazeera) hospital
Locations (1):
- Aljazeera (Al Gazeera) hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No